CLINICAL TRIAL: NCT05430919
Title: A Two-Part Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy of the Anti-Bet v 1 Monoclonal Antibodies to Reduce Allergic Rhinitis and Conjunctivitis Symptoms and Skin Test Reactivity Upon Exposure to Birch Allergen
Brief Title: Efficacy of the Anti-Bet v 1 Monoclonal Antibodies (Given Subcutaneously) to Reduce Allergic Rhinitis and Conjunctivitis Symptoms and Skin Test Reactivity Upon Exposure to Birch Allergen in Adult Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R5713-5714-5715-ALG-21111
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Allergic Rhinitis; Conjunctivitis
Keywords: Birch Allergy; Birch Pollen Season; Monoclonal antibody(ies); Oak Pollen Season; Subcutaneous immunotherapy; Skin Prick Test
MeSH Terms: conditions — Rhinitis, Allergic; Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- REGN5713-5714-5715 (Experimental): 3-mAb
  Interventions: Drug: REGN5713; Drug: REGN5714; Drug: REGN5715
- REGN5713-5715 (Experimental): 2-mAb
  Interventions: Drug: REGN5713; Drug: REGN5715; Other: Placebo
- REGN5715 (Experimental): 1-mAb
  Interventions: Drug: REGN5715; Other: Placebo
- Matching Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: REGN5713 — Administered subcutaneously (SC)
  Arms: REGN5713-5714-5715; REGN5713-5715
Drug: REGN5714 — Administered SC
  Arms: REGN5713-5714-5715
Drug: REGN5715 — Administered SC
  Arms: REGN5713-5714-5715; REGN5713-5715; REGN5715
Other: Placebo — Administered SC
  Arms: Matching Placebo; REGN5713-5715; REGN5715

SUMMARY:
Primary objective: To assess the efficacy of a single dose of the anti- Bet v 1 monoclonal antibodies (mAb(s ) in the reduction of allergic nasal symptoms during an out-of-season birch allergen environmental exposure unit (EEU) challenge in participants receiving REGN5713-5714-5715 versus placebo (Part A)

DETAILED DESCRIPTION:
The study consists of Part A and Part B. All participants will be asked to complete both Part A and Part B of the study. The study lasts for a total duration of up to approximately 46 weeks (including up to a 10-week screening period). Part A of the study lasts up to approximately 28 weeks (including the screening period). Part B of the study starts after completion of Part A and lasts up to approximately 18 weeks (including an approximately 4-week follow-up period after end of birch pollen season (BPS)), dependent on the start and end times of the natural BPS.

ELIGIBILITY:
Key Inclusion Criteria:

1. Documented or participant-reported history of birch tree pollen-triggered allergic-rhinitis (AR) symptoms with or without conjunctivitis (for at least 2 seasons)
2. Positive Skin prick test (SPT) with birch tree pollen extract (mean wheal diameter at least 5 mm greater than a negative control) in screening period
3. Positive allergen-specific immunoglobulin E (sIgE) tests for birch tree pollen and Bet v 1 (≥0.7 kUa/L) in screening period
4. Demonstrated TNSS ≥ 6 out of 12 on at least 2 time points during the birch EEU exposure challenge in screening period

Key Exclusion Criteria:

1. Participation in a prior REGN5713-5714-5715 clinical trial and received REGN5713-5714-5715 antibodies (receipt of placebo in a previous trial is allowed)
2. Significant rhinitis, sinusitis, significant and/or severe allergies not associated with the birch pollen season, or due to daily contact with other non-birch related allergens causing symptoms that are expected to coincide or potentially interfere with the study EEU assessments or with the birch pollen season, as assessed by the investigator
3. Participants who anticipate major changes in allergen exposure during the birch pollen season that are expected to coincide with study assessments or planned travel that is expected to interfere with the study assessments, as assessed by the investigator (eg. anticipated travel during planned EEU sessions or birch pollen season)
4. Persistent chronic or recurring acute infection requiring treatment with antibiotics, antivirals, or antifungals, or any untreated respiratory infections within 4 weeks prior to screening visit 1. Patients may be re-evaluated for eligibility after resolution of symptoms and specified duration.
5. History of significant, recurrent sinusitis, defined as at least 3 episodes requiring antibiotic treatment per year for the last 2 years
6. Abnormal lung function as judged by the investigator with Forced Expiratory Volume (FEV1) <75% of predicted at screening or randomization
7. A clinical history of moderate to severe asthma, uncontrolled asthma, global initiative for asthma [GINA] steps 3 to 5, history of life-threatening asthma, asthma exacerbations due to tree pollen allergy within 2 prior seasons, >2 asthma exacerbations requiring systemic steroids in past 12 months, asthma related emergency care or hospitalization within 12 months prior to screening, as defined in the protocol.
8. History of birch or other tree allergen immunotherapy in the 3 years prior to screening.
9. Use of anti-IgE or other biological therapy (including but not limited to anti IL-5, anti IL-4) that interferes with type 2 disease within 6 months prior to screening visit 1.
10. Allergen-specific immunotherapy with any allergen other than birch or other trees at screening.
11. History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric, or neurological disease,
12. Any malignancy within the past 5 years, except for basal cell or squamous epithelial cell carcinomas of the skin or carcinoma in situ of the cervix or anus that have been resected, with no evidence of local recurrence or metastatic disease for 3 years.

NOTE: Other protocol defined Inclusion/Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (3):
- Canada (3):
  - Kingston General Health Research Institute, Kingston, Ontario
  - Inflamax Research Limited DBA Cliantha Research, Mississauga, Ontario
  - Clinique Specialisee en Allergie de la Capitale, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual anonymized participant data will be considered for sharing once the indication has been approved by a regulatory body, if there is legal authority to share the data and there is not a reasonable likelihood of participant re-identification.
Access Criteria: Qualified researchers may request access to anonymized patient level data or aggregate study data when Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency [EMA], Pharmaceuticals and Medical Devices Agency [PMDA], etc) for the product and indication, has the legal authority to share the data, and has made the study results publicly available (eg, scientific publication, scientific conference, clinical trial registry).
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 847 participants were screened, of which 217 were randomized
Groups:
- Placebo: Matching placebo
- REGN5715 300 mg: 1-monoclonal antibody (mAb) REGN5715 300 mg plus placebo to replace REGN5713-5714
- REGN5713-5715 600 mg: 2-monoclonal antibody (mAb) cocktail REGN5713-5715 600 mg (300 mg per mAb) plus placebo to replace REGN5714
- REGN5713-5714-5715 900 mg: 3-monoclonal antibody (mAb) cocktail REGN5713-5714-5715 900 mg (300 mg per mAb)
Period: Overall Study
Arm/Group | Placebo | REGN5715 300 mg | REGN5713-5715 600 mg | REGN5713-5714-5715 900 mg
Started | 55 | 55 | 52 | 55
Completed | 52 | 54 | 51 | 54
Not Completed | 3 | 1 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | REGN5715 300 mg | REGN5713-5715 600 mg | REGN5713-5714-5715 900 mg | Total
Number analyzed (Participants) | 55 | 55 | 52 | 55 | 217
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.8 (13.72) | 40.1 (11.15) | 40.3 (10.87) | 42.6 (12.56) | 41.7 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 27 | 22 | 34 | 113
  Male | 25 | 28 | 30 | 21 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 6 | 5 | 21
  Not Hispanic or Latino | 49 | 47 | 46 | 49 | 191
  Unknown or Not Reported | 1 | 3 | 0 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 7 | 6 | 8 | 12 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 5 | 5 | 21
  White | 39 | 43 | 37 | 36 | 155
  More than one race | 1 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 2 | 0 | 1 | 2 | 5
Birch allergen EEU Mean Total Nasal Symptom Score (TNSS) (0 - 12) (2-6 Hours) [Mean (Standard Deviation); unit: Scores on a Scale] — Mean TNSS (0 - 12) (2 to 6 hours) during a birch allergen environmental exposure unit (EEU) challenge. The TNSS ranges from 0 to 12 and is based on assessment of 4 nasal symptoms graded on a Likert scale ranging from 0 (none) to 3 (severe) for nasal congestion, itching, and runny nose, and sneezing. Higher score indicates worse outcome.
  Scores on a Scale | 7.36 (2.489) | 7.84 (2.479) | 7.29 (2.414) | 7.71 (2.549) | 7.55 (2.477)

OUTCOME MEASURES:

1. Primary Outcome: Mean Total Nasal Symptom Score (TNSS) (2 to 6 Hours) During Out-of-season Birch Allergen Environmental Exposure Unit (EEU) Challenge (REGN5713-5714-5715 vs. Placebo) at Day 29
Description: TNSS ranges from 0 (none) to 12 (severe): sum of 4 nasal symptoms (nasal congestion, itching, & runny nose, & sneezing) graded on a Likert scale ranging from 0 (none) to 3 (severe); Higher score indicates worse outcome.
Time Frame: Day 29 from randomization (Out-of-season)
Population: Randomized participants in only the REGN5713-5714-5715 and placebo arms were assessed for this endpoint. Missing values were imputed using multiple imputation (MI) method.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 900 mg | Placebo
Number analyzed (Participants) | 55 | 55
Scores on a Scale | 4.40 (0.377) | 6.71 (0.380)
Statistical Analysis 1: Comparison: REGN5713-5714-5715 900 mg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares (LS) Mean Difference = -2.31, 95% CI 2-sided [-3.229 to -1.385] — REGN5713-5714-5715 900 mg vs. Placebo, Day 29

2. Secondary Outcome: Mean TNSS (2 to 6 Hours) During Out-of-season Birch Allergen EEU Challenge (Except for REGN5713-5714-5715) at Day 29
Description: as for outcome 1
Time Frame: Day 29 from randomization (Out-of-season)
Population: Randomized participants in only the REGN5713-5715, REGN5715 and placebo arms were assessed for this endpoint. Missing values were imputed using multiple imputation (MI) method.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 52 | 55 | 55
Scores on a Scale | 4.06 (0.406) | 5.20 (0.393) | 6.71 (0.380)
Statistical Analysis 1: Comparison: REGN5713-5715 600 mg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -2.65, 95% CI 2-sided [-3.634 to -1.658] — REGN5713-5715 600 mg vs. Placebo, Day 29
Statistical Analysis 2: Comparison: REGN5715 300 mg vs Placebo; Test type: Superiority; p = 0.0023, ANCOVA; LS Mean Difference = -1.51, 95% CI 2-sided [-2.478 to -0.539] — REGN5715 300 mg vs. Placebo, Day 29

3. Secondary Outcome: Mean TNSS (2 to 6 Hours) During Out-of-season Birch Allergen EEU Challenge at Day 57 and Day 85
Description: as for outcome 1
Time Frame: Day 57 and Day 85, from randomization (Out-of-season)
Population: The overall "Number of Participants Analyzed" is the total number of randomized participants in each treatment group. The "Number Analyzed" for each timepoint is the number of participants with available observed data that were analyzed at that timepoint.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 55 | 52 | 55 | 55
Scores on a Scale
  Day 57: number analyzed (Participants) | 43 | 40 | 44 | 42
  Day 57 | 4.47 (0.458) | 3.89 (0.471) | 5.58 (0.451) | 6.29 (0.445)
  Day 85: number analyzed (Participants) | 37 | 38 | 40 | 41
  Day 85 | 4.61 (0.511) | 4.48 (0.506) | 5.38 (0.499) | 6.14 (0.466)

4. Secondary Outcome: Mean Total Ocular Symptom Score (TOSS) (2 to 6 Hours) During Out-of-season Birch Allergen EEU Challenge at Day 29
Description: TOSS ranges from 0 (none) to 6 (severe): sum of 2 eye symptoms graded on a Likert scale each ranging from 0 (none) to 3 (severe) for itching/redness/gritty feeling & tearing/watering; Higher score indicates worse outcome.
Time Frame: Day 29 from randomization (Out-of-season)
Population: All randomized participants. Missing values were imputed using multiple imputation (MI) method.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 55 | 52 | 55 | 55
Scores on a Scale | 1.81 (0.202) | 1.69 (0.217) | 2.01 (0.207) | 2.48 (0.202)

5. Secondary Outcome: Mean TOSS (2 to 6 Hours) During Out-of-season Birch Allergen EEU Challenge at Day 57 and Day 85
Description: as for outcome 4
Time Frame: Day 57 and Day 85, from randomization (Out-of-season)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 55 | 52 | 55 | 55
Scores on a Scale
  Day 57: number analyzed (Participants) | 43 | 40 | 44 | 42
  Day 57 | 1.63 (0.231) | 1.66 (0.237) | 2.04 (0.227) | 2.57 (0.225)
  Day 85: number analyzed (Participants) | 37 | 38 | 40 | 41
  Day 85 | 1.90 (0.243) | 1.96 (0.241) | 1.91 (0.238) | 2.51 (0.223)

6. Secondary Outcome: Mean Total Symptom Score (TSS) (2 to 6 Hours) During Out-of-season Birch Allergen EEU Challenge at Day 29
Description: TSS ranges from 0 (none) to 18 (severe): sum of TNSS & TOSS combined; Higher score indicates worse outcome
Time Frame: Day 29 from randomization (Out-of-season)
Population: All randomized participants. Missing values were imputed using multiple imputation (MI) method.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 55 | 52 | 55 | 55
Scores on a Scale | 6.22 (0.549) | 5.76 (0.592) | 7.21 (0.572) | 9.20 (0.553)

7. Secondary Outcome: Mean TSS (2 to 6 Hours) During Out-of-season Birch Allergen EEU Challenge at Day 57 and at Day 85
Description: TSS ranges from 0 (none) to 18 (severe): sum of TNSS & TOSS combined; Higher score indicates worse outcome
Time Frame: Day 57 and Day 85, from randomization (Out-of-season)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 55 | 52 | 55 | 55
Scores on a Scale
  Day 57: number analyzed (Participants) | 43 | 40 | 44 | 42
  Day 57 | 6.09 (0.652) | 5.57 (0.671) | 7.62 (0.642) | 8.86 (0.634)
  Day 85: number analyzed (Participants) | 37 | 38 | 40 | 41
  Day 85 | 6.49 (0.710) | 6.44 (0.703) | 7.30 (0.693) | 8.63 (0.648)

8. Secondary Outcome: Change From Pre-treatment Baseline in TNSS (2 to 6 Hours) During Out-of-season Birch Allergen EEU Challenge at Days 29, 57 and 85
Description: as for outcome 1
Time Frame: Day 29, Day 57 and Day 85, from randomization (Out-of-season)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 55 | 52 | 55 | 55
Scores on a Scale
  Day 29: number analyzed (Participants) | 51 | 40 | 49 | 48
  Day 29 | -3.14 (0.371) | -3.52 (0.411) | -2.27 (0.373) | -0.84 (0.376)
  Day 57: number analyzed (Participants) | 43 | 40 | 44 | 42
  Day 57 | -3.14 (0.458) | -3.71 (0.471) | -2.03 (0.451) | -1.31 (0.445)
  Day 85: number analyzed (Participants) | 37 | 38 | 40 | 41
  Day 85 | -3.04 (0.511) | -3.17 (0.506) | -2.27 (0.499) | -1.50 (0.466)

9. Secondary Outcome: Change From Pre-treatment Baseline in TOSS (2 to 6 Hours) During Out-of-season Birch Allergen EEU Challenge at Days 29, 57 and 85
Description: as for outcome 4
Time Frame: Day 29, Day 57 and Day 85, from randomization (Out-of-season)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 55 | 52 | 55 | 55
Scores on a Scale
  Day 29: number analyzed (Participants) | 51 | 40 | 49 | 48
  Day 29 | -1.11 (0.202) | -1.26 (0.222) | -0.87 (0.202) | -0.44 (0.204)
  Day 57: number analyzed (Participants) | 43 | 40 | 44 | 42
  Day 57 | -1.41 (0.231) | -1.37 (0.237) | -100 (0.227) | -0.47 (0.225)
  Day 85: number analyzed (Participants) | 37 | 38 | 40 | 41
  Day 85 | -1.15 (0.243) | -1.09 (0.241) | -1.14 (0.238) | -0.54 (0.223)

10. Secondary Outcome: Change From Pre-treatment Baseline in TSS (2 to 6 Hours) During Out-of-season Birch Allergen EEU Challenge at Days 29, 57 and 85
Description: TSS ranges from 0 (none) to 18 (severe): sum of TNSS & TOSS combined; Higher score indicates worse outcome
Time Frame: Day 29, Day 57 and Day 85, from randomization (Out-of-season)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 55 | 52 | 55 | 55
Scores on a Scale
  Day 29: number analyzed (Participants) | 51 | 40 | 49 | 48
  Day 29 | -4.24 (0.543) | -4.76 (0.600) | -3.14 (0.545) | -1.26 (0.550)
  Day 57: number analyzed (Participants) | 43 | 40 | 44 | 42
  Day 57 | -4.55 (0.652) | -5.08 (0.671) | -3.02 (0.642) | -1.78 (0.634)
  Day 85: number analyzed (Participants) | 37 | 38 | 40 | 41
  Day 85 | -4.20 (0.710) | -4.26 (0.703) | -3.39 (0.693) | -2.06 (0.648)

11. Secondary Outcome: Percent Change From Pre-treatment Baseline in TNSS (2 to 6 Hours) During Out-of-season Birch Allergen EEU Challenge at Days 29, 57 and 85
Description: as for outcome 1
Time Frame: Day 29, Day 57 and Day 85, from randomization (Out-of-season)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percentage of Change
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 55 | 52 | 55 | 55
Percentage of Change
  Day 29: number analyzed (Participants) | 51 | 40 | 49 | 48
  Day 29 | -44.35 (5.099) | -46.86 (5.645) | -27.88 (5.132) | -4.10 (5.173)
  Day 57: number analyzed (Participants) | 53 | 40 | 44 | 42
  Day 57 | -42.98 (6.508) | -48.26 (6.689) | -29.48 (6.407) | -11.65 (6.318)
  Day 85: number analyzed (Participants) | 37 | 38 | 40 | 41
  Day 85 | -41.94 (7.683) | -39.22 (7.607) | -28.94 (7.505) | -13.99 (7.003)

12. Secondary Outcome: Percent Change From Pre-treatment Baseline in TOSS (2 to 6 Hours) During Out-of-season Birch Allergen EEU Challenge at Days 29, 57 and 85
Description: as for outcome 4
Time Frame: Day 29, Day 57 and Day 85, from randomization (Out-of-season)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percentage of Change
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 55 | 52 | 55 | 55
Percentage of Change
  Day 29: number analyzed (Participants) | 51 | 40 | 49 | 48
  Day 29 | -44.15 (7.729) | -40.40 (8.504) | -29.90 (7.731) | -8.40 (7.807)
  Day 57: number analyzed (Participants) | 43 | 40 | 44 | 42
  Day 57 | -53.08 (7.932) | -44.70 (8.147) | -35.02 (7.795) | -11.64 (7.725)
  Day 85: number analyzed (Participants) | 37 | 38 | 40 | 41
  Day 85 | -46.38 (9.206) | -32.54 (9.117) | -39.16 (8.997) | -12.17 (8.431)

13. Secondary Outcome: Percent Change From Pre-treatment Baseline in TSS (2 to 6 Hours) During Out-of-season Birch Allergen EEU Challenge at Days 29, 57 and Day 85
Description: TSS ranges from 0 (none) to 18 (severe): sum of TNSS & TOSS combined; Higher score indicates worse outcome
Time Frame: Day 29, Day 57 and Day 85, from randomization (Out-of-season)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percentage of Change
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 55 | 52 | 55 | 55
Percentage of Change
  Day 29: number analyzed (Participants) | 51 | 40 | 49 | 48
  Day 29 | -44.33 (5.274) | -44.97 (5.830) | -27.50 (5.298) | -4.18 (5.347)
  Day 57: number analyzed (Participants) | 43 | 40 | 44 | 42
  Day 57 | -45.49 (6.283) | -46.81 (6.460) | -30.21 (6.182) | -10.55 (6.110)
  Day 85: number analyzed (Participants) | 37 | 38 | 40 | 41
  Day 85 | 42.74 (7.252) | -37.11 (7.186) | -31.64 (7.084) | -13.55 (6.621)

14. Secondary Outcome: Change From Pre-treatment Baseline in the Birch Titrated Skin Prick Test (SPT) Mean Wheal Diameter Area Under the Curve (AUC) at Day 29
Description: Titrated skin prick test (SPT) AUC= The skin prick test mean wheal diameters [mm] using serial dilutions of the allergen were used to calculate an AUC. AUC of titrated SPT mean wheal diameters were derived using the trapezoidal rule. For each participant, the AUC was calculated for the mean wheal diameter calculated over titrated concentrations of the allergen on a log scale and then normalized.
Time Frame: Day 29 from randomization (Out-of-season)
Population: All randomized participants
Measure: Least Squares Mean (Standard Error); unit: millimeter (mm)
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 55 | 52 | 55 | 55
millimeter (mm) | -5.396 (0.2822) | -4.743 (0.3243) | -3.266 (0.2983) | -0.507 (0.2946)

15. Secondary Outcome: Change From Pre-treatment Baseline in the Birch Titrated SPT Mean Wheal Diameter AUC at Day 57 and Day 85
Description: as for outcome 14
Time Frame: Day 57 and Day 85, from randomization (Out-of-season)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: millimeter (mm)
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 55 | 52 | 55 | 55
millimeter (mm)
  Day 57: number analyzed (Participants) | 43 | 40 | 44 | 42
  Day 57 | -5.110 (0.2878) | -4.693 (0.2976) | -3.052 (0.2837) | -0.054 (0.2789)
  Day 85: number analyzed (Participants) | 37 | 38 | 40 | 41
  Day 85 | -4.418 (0.3218) | -4.241 (0.3199) | -1.757 (0.3166) | 0.016 (0.2930)

16. Secondary Outcome: Change From Pre-treatment Baseline in the Birch Titrated SPT Mean Wheal Diameter AUC at Day 127
Description: as for outcome 14
Time Frame: Day 127 from randomization
Population: Randomized participants with Day 127 visit (intended to be pre-season) at least 12 weeks post-randomization
Measure: Least Squares Mean (Standard Error); unit: millimeter (mm)
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 28 | 26 | 31 | 31
millimeter (mm) | -3.980 (0.3673) | -3.590 (0.3907) | -2.485 (0.3539) | 0.058 (0.3481)

17. Secondary Outcome: Change From Pre-treatment Baseline in the Birch Titrated SPT Mean Wheal Diameter AUC at Day 225 and Day 253
Description: as for outcome 14
Time Frame: Day 225 from randomization (end-of-season) and Day 253 from randomization (end of study)
Population: Among randomized participants that received a second dose of study drug, the number of participants analyzed is the number of participants with a baseline measurement and post-baseline measurement. The number analyzed for each timepoint is the number of participants with available observed data that were analyzed at that timepoint.
Measure: Least Squares Mean (Standard Error); unit: millimeter (mm)
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 38 | 33 | 39 | 39
millimeter (mm)
  Day 225: number analyzed (Participants) | 27 | 15 | 22 | 21
  Day 225 | -5.435 (0.3648) | -4.587 (0.4578) | -3.263 (0.3983) | -0.715 (0.3984)
  Day 253: number analyzed (Participants) | 38 | 33 | 39 | 38
  Day 253 | -4.752 (0.3184) | -4.546 (0.3329) | -2.802 (0.3113) | -0.759 (0.3007)

18. Secondary Outcome: Percent Change From Pre-treatment Baseline in the Birch Titrated SPT Mean Wheal Diameter AUC at Day 29
Description: as for outcome 14
Time Frame: Day 29 from randomization (Out-of-season)
Population: All randomized participants
Measure: Least Squares Mean (Standard Error); unit: Percentage of Change
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 55 | 52 | 55 | 55
Percentage of Change | -66.50 (4.036) | -59.32 (4.689) | -38.14 (4.217) | -3.31 (4.223)
Statistical Analysis 1: Comparison: REGN5713-5714-5715 900 mg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -63.18, 95% CI 2-sided [-73.411 to -52.950] — REGN5713-5714-5715 900 mg vs. Placebo, Day 29
Statistical Analysis 2: Comparison: REGN5713-5715 600 mg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -56.01, 95% CI 2-sided [-66.806 to -45.204] — REGN5713-5715 600 mg vs. Placebo, Day 29
Statistical Analysis 3: Comparison: REGN5715 300 mg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; LS Mean Difference = -34.82, 95% CI 2-sided [-45.304 to -24.343] — REGN5715 300 mg vs. Placebo, Day 29

19. Secondary Outcome: Percent Change From Pre-treatment Baseline in the Birch Titrated SPT Mean Wheal Diameter AUC at Day 57 and Day 85
Description: as for outcome 14
Time Frame: Day 57 and Day 85, from randomization (Out-of-season)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percentage of Change
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 55 | 52 | 55 | 55
Percentage of Change
  Day 57: number analyzed (Participants) | 43 | 40 | 44 | 42
  Day 57 | -64.45 (4.917) | -59.19 (5.084) | -37.04 (4.847) | 8.07 (4.765)
  Day 85: number analyzed (Participants) | 37 | 38 | 40 | 41
  Day 85 | -54.36 (5.108) | -54.43 (5.079) | -18.38 (5.026) | 7.85 (4.651)

20. Secondary Outcome: Percent Change From Pre-treatment Baseline in the Birch Titrated SPT Mean Wheal Diameter AUC at Day 127
Description: as for outcome 14
Time Frame: Day 127 from randomization
Population: Randomized participants with Day 127 visit (intended to be pre-season) at least 12 weeks post-randomization
Measure: Least Squares Mean (Standard Error); unit: Percentage of Change
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 28 | 26 | 31 | 31
Percentage of Change | -49.10 (5.715) | -44.38 (6.079) | -29.13 (5.506) | 9.30 (5.416)

21. Secondary Outcome: Percent Change From Pre-treatment Baseline in the Birch Titrated SPT Mean Wheal Diameter AUC at Day 225 and Day 253
Description: as for outcome 14
Time Frame: Day 225 from randomization (end-of-season) and Day 253 from randomization (end of study)
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: Percentage of Change
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 38 | 33 | 39 | 39
Percentage of Change
  Day 225: number analyzed (Participants) | 27 | 15 | 22 | 21
  Day 225 | -72.42 (5.621) | -57.83 (7.054) | -36.74 (6.136) | -6.70 (6.138)
  Day 253: number analyzed (Participants) | 38 | 33 | 39 | 38
  Day 253 | -62.71 (5.010) | -60.89 (5.238) | -30.98 (4.898) | -5.41 (4.732)

22. Secondary Outcome: Mean TNSS, TOSS and TSS (2 to 6 Hours) During Out-of-season Oak Allergen EEU Challenge at Day 36
Description: TNSS ranges from 0 (none) to 12 (severe): sum of 4 nasal symptoms (nasal congestion, itching, & runny nose, & sneezing) graded on a Likert scale ranging from 0 (none) to 3 (severe); Higher score indicates worse outcome. TOSS ranges from 0 (none) to 6 (severe): sum of 2 eye symptoms graded on a Likert scale each ranging from 0 (none) to 3 (severe) for itching/redness/gritty feeling & tearing/watering; Higher score indicates worse outcome. TSS ranges from 0 (none) to 18 (severe): sum of TNSS & TOSS combined; Higher score indicates worse outcome.
Time Frame: Day 36 from randomization (Out-of-season)
Population: The "Number of Participants Analyzed" is the number of participants allergic to oak with a baseline measurement and post-baseline measurement in each treatment group. The "Number Analyzed" for each scale is the number of participants with available observed data for that scale.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 29 | 28 | 35 | 30
Scores on a Scale
  TNSS | 4.79 (0.561) | 4.53 (0.570) | 5.04 (0.516) | 5.59 (0.538)
  TOSS | 1.86 (0.280) | 2.05 (0.284) | 1.78 (0.256) | 2.54 (0.270)
  TSS | 6.64 (0.804) | 6.57 (0.817) | 6.82 (0.738) | 8.08 (0.771)

23. Secondary Outcome: Change From Pre-treatment Baseline in TNSS, TOSS and TSS (2 to 6 Hours) During Oak Allergen EEU Challenge at Day 36
Description: as for outcome 22
Time Frame: Day 36 from randomization (Out-of-season)
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 29 | 28 | 35 | 30
Scores on a Scale
  TNSS | -2.63 (0.561) | -2.89 (0.570) | -2.38 (0.516) | -1.83 (0.538)
  TOSS | -1.33 (0.280) | -1.14 (0.284) | -1.41 (0.256) | -0.65 (0.270)
  TSS | -3.97 (0.804) | -4.04 (0.817) | -3.79 (0.738) | -2.53 (0.771)

24. Secondary Outcome: Percent Change From Pre-treatment Baseline in TNSS, TOSS and TSS (2 to 6 Hours) During Oak Allergen EEU Challenge at Day 36
Description: as for outcome 22
Time Frame: Day 36 from randomization (Out-of-season)
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: Percentage of Change
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 29 | 28 | 35 | 30
Percentage of Change
  TNSS | -35.18 (7.448) | -34.95 (7.572) | -30.36 (6.848) | -20.46 (7.144)
  TOSS | -52.74 (9.947) | -32.95 (10.097) | -49.39 (9.113) | -15.45 (9.589)
  TSS | -38.98 (7.471) | -33.81 (7.590) | -35.14 (6.858) | -19.25 (7.167)

25. Secondary Outcome: Number of Participants Achieving Different Degrees of Clinical Responses Compared Across TNSS (2 to 6 Hours) Response Thresholds
Description: as for outcome 1
Time Frame: Day 29, Day 57 and Day 85, from randomization (Out-of-season)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | REGN5715 300 mg | REGN5713-5715 600 mg | REGN5713-5714-5715 900 mg
Number analyzed (Participants) | 55 | 55 | 52 | 55
Participants
  Day 29 Participants with a percent reduction of at least 75% or greater: number analyzed (Participants) | 48 | 49 | 40 | 51
  Day 29 Participants with a percent reduction of at least 75% or greater | 2 | 1 | 11 | 9
  Day 29 Participants with a percent reduction of at least 50% or greater: number analyzed (Participants) | 48 | 49 | 40 | 51
  Day 29 Participants with a percent reduction of at least 50% or greater | 7 | 13 | 23 | 23
  Day 29 Participants with a percent reduction of at least 25% or greater: number analyzed (Participants) | 48 | 49 | 40 | 51
  Day 29 Participants with a percent reduction of at least 25% or greater | 13 | 31 | 31 | 40
  Day 57 Participants with a percent reduction of at least 75% or greater: number analyzed (Participants) | 42 | 44 | 40 | 43
  Day 57 Participants with a percent reduction of at least 75% or greater | 3 | 6 | 13 | 6
  Day 57 Participants with a percent reduction of at least 50% or greater: number analyzed (Participants) | 42 | 44 | 40 | 43
  Day 57 Participants with a percent reduction of at least 50% or greater | 7 | 14 | 21 | 17
  Day 57 Participants with a percent reduction of at least 25% or greater: number analyzed (Participants) | 42 | 44 | 40 | 43
  Day 57 Participants with a percent reduction of at least 25% or greater | 15 | 27 | 30 | 31
  Day 85 Participants with a percent reduction of at least 75% or greater: number analyzed (Participants) | 41 | 40 | 38 | 37
  Day 85 Participants with a percent reduction of at least 75% or greater | 4 | 7 | 10 | 7
  Day 85 Participants with a percent reduction of at least 50% or greater: number analyzed (Participants) | 41 | 40 | 38 | 37
  Day 85 Participants with a percent reduction of at least 50% or greater | 9 | 15 | 18 | 15
  Day 85 Participants with a percent reduction of at least 25% or greater: number analyzed (Participants) | 41 | 40 | 38 | 37
  Day 85 Participants with a percent reduction of at least 25% or greater | 17 | 26 | 26 | 30

26. Secondary Outcome: Number of Participants Achieving Different Degrees of Clinical Responses Compared Across TOSS (2 to 6 Hours) Response Thresholds
Description: as for outcome 4
Time Frame: Day 29, Day 57 and Day 85, from randomization (Out-of-season)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | REGN5715 300 mg | REGN5713-5715 600 mg | REGN5713-5714-5715 900 mg
Number analyzed (Participants) | 55 | 55 | 52 | 55
Participants
  Day 29 Participants with a percent reduction of at least 75% or greater: number analyzed (Participants) | 48 | 49 | 40 | 51
  Day 29 Participants with a percent reduction of at least 75% or greater | 8 | 6 | 12 | 16
  Day 29 Participants with a percent reduction of at least 50% or greater: number analyzed (Participants) | 48 | 49 | 40 | 51
  Day 29 Participants with a percent reduction of at least 50% or greater | 10 | 18 | 20 | 28
  Day 29 Participants with a percent reduction of at least 25% or greater: number analyzed (Participants) | 48 | 49 | 40 | 51
  Day 29 Participants with a percent reduction of at least 25% or greater | 22 | 34 | 29 | 38
  Day 57 Participants with a percent reduction of at least 75% or greater: number analyzed (Participants) | 42 | 44 | 40 | 43
  Day 57 Participants with a percent reduction of at least 75% or greater | 7 | 10 | 20 | 20
  Day 57 Participants with a percent reduction of at least 50% or greater: number analyzed (Participants) | 42 | 44 | 40 | 43
  Day 57 Participants with a percent reduction of at least 50% or greater | 9 | 22 | 25 | 27
  Day 57 Participants with a percent reduction of at least 25% or greater: number analyzed (Participants) | 42 | 44 | 40 | 43
  Day 57 Participants with a percent reduction of at least 25% or greater | 17 | 26 | 26 | 31
  Day 85 Participants with a percent reduction of at least 75% or greater: number analyzed (Participants) | 41 | 40 | 38 | 37
  Day 85 Participants with a percent reduction of at least 75% or greater | 5 | 10 | 14 | 11
  Day 85 Participants with a percent reduction of at least 50% or greater: number analyzed (Participants) | 41 | 40 | 38 | 37
  Day 85 Participants with a percent reduction of at least 50% or greater | 13 | 21 | 19 | 20
  Day 85 Participants with a percent reduction of at least 25% or greater: number analyzed (Participants) | 41 | 40 | 38 | 37
  Day 85 Participants with a percent reduction of at least 25% or greater | 18 | 30 | 24 | 30

27. Secondary Outcome: Number of Participants Achieving Different Degrees of Clinical Responses Compared Across TSS (2 to 6 Hours) Response Thresholds
Description: TSS ranges from 0 (none) to 18 (severe): sum of TNSS & TOSS combined; Higher score indicates worse outcome.
Time Frame: Day 29, Day 57 and Day 85, from randomization (Out-of-season)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | REGN5715 300 mg | REGN5713-5715 600 mg | REGN5713-5714-5715 900 mg
Number analyzed (Participants) | 55 | 55 | 52 | 55
Participants
  Day 29 Participants with a percent reduction of at least 75% or greater: number analyzed (Participants) | 48 | 49 | 40 | 51
  Day 29 Participants with a percent reduction of at least 75% or greater | 3 | 2 | 11 | 11
  Day 29 Participants with a percent reduction of at least 50% or greater: number analyzed (Participants) | 48 | 49 | 40 | 51
  Day 29 Participants with a percent reduction of at least 50% or greater | 7 | 13 | 23 | 21
  Day 29 Participants with a percent reduction of at least 25% or greater: number analyzed (Participants) | 48 | 49 | 40 | 51
  Day 29 Participants with a percent reduction of at least 25% or greater | 13 | 30 | 29 | 40
  Day 57 Participants with a percent reduction of at least 75% or greater: number analyzed (Participants) | 42 | 44 | 40 | 43
  Day 57 Participants with a percent reduction of at least 75% or greater | 3 | 4 | 14 | 9
  Day 57 Participants with a percent reduction of at least 50% or greater: number analyzed (Participants) | 42 | 44 | 40 | 43
  Day 57 Participants with a percent reduction of at least 50% or greater | 7 | 15 | 23 | 22
  Day 57 Participants with a percent reduction of at least 25% or greater: number analyzed (Participants) | 42 | 44 | 40 | 43
  Day 57 Participants with a percent reduction of at least 25% or greater | 15 | 25 | 29 | 32
  Day 85 Participants with a percent reduction of at least 75% or greater: number analyzed (Participants) | 41 | 40 | 38 | 37
  Day 85 Participants with a percent reduction of at least 75% or greater | 4 | 7 | 8 | 8
  Day 85 Participants with a percent reduction of at least 50% or greater: number analyzed (Participants) | 41 | 40 | 38 | 37
  Day 85 Participants with a percent reduction of at least 50% or greater | 8 | 14 | 18 | 16
  Day 85 Participants with a percent reduction of at least 25% or greater: number analyzed (Participants) | 41 | 40 | 38 | 37
  Day 85 Participants with a percent reduction of at least 25% or greater | 18 | 29 | 25 | 32

28. Secondary Outcome: Number of Participants Achieving Different Degrees of Responses in the Birch Titrated SPT Mean Wheal Diameter AUC Compared Across Different Response Thresholds
Description: as for outcome 14
Time Frame: Day 29, Day 57 and Day 85, from randomization (Out-of-season)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | REGN5715 300 mg | REGN5713-5715 600 mg | REGN5713-5714-5715 900 mg
Number analyzed (Participants) | 55 | 55 | 52 | 55
Participants
  Day 29 Participants with a percent reduction of at least 75% or greater: number analyzed (Participants) | 48 | 50 | 41 | 53
  Day 29 Participants with a percent reduction of at least 75% or greater | 1 | 1 | 8 | 19
  Day 29 Participants with a percent reduction of at least 50% or greater: number analyzed (Participants) | 48 | 50 | 41 | 53
  Day 29 Participants with a percent reduction of at least 50% or greater | 1 | 12 | 24 | 41
  Day 29 Participants with a percent reduction of at least 25% or greater: number analyzed (Participants) | 48 | 50 | 41 | 53
  Day 29 Participants with a percent reduction of at least 25% or greater | 11 | 34 | 35 | 50
  Day 57 Participants with a percent reduction of at least 75% or greater: number analyzed (Participants) | 42 | 44 | 40 | 43
  Day 57 Participants with a percent reduction of at least 75% or greater | 0 | 1 | 4 | 12
  Day 57 Participants with a percent reduction of at least 50% or greater: number analyzed (Participants) | 42 | 44 | 40 | 43
  Day 57 Participants with a percent reduction of at least 50% or greater | 1 | 9 | 27 | 25
  Day 57 Participants with a percent reduction of at least 25% or greater: number analyzed (Participants) | 42 | 44 | 40 | 43
  Day 57 Participants with a percent reduction of at least 25% or greater | 5 | 29 | 34 | 40
  Day 85 Participants with a percent reduction of at least 75% or greater: number analyzed (Participants) | 41 | 40 | 38 | 37
  Day 85 Participants with a percent reduction of at least 75% or greater | 0 | 0 | 11 | 8
  Day 85 Participants with a percent reduction of at least 50% or greater: number analyzed (Participants) | 41 | 40 | 38 | 37
  Day 85 Participants with a percent reduction of at least 50% or greater | 1 | 2 | 21 | 25
  Day 85 Participants with a percent reduction of at least 25% or greater: number analyzed (Participants) | 41 | 40 | 38 | 37
  Day 85 Participants with a percent reduction of at least 25% or greater | 5 | 17 | 31 | 32

29. Secondary Outcome: Mean TNSS, TOSS and TSS (2 to 6 Hours) During Peak-season Birch Allergen EEU Challenge at Day 190
Description: Peak season EEU is an in-season challenge corresponding to approximate timing of the anticipated peak BPS; TNSS ranges from 0 (none) to 12 (severe): sum of 4 nasal symptoms (nasal congestion, itching, & runny nose, & sneezing) graded on a Likert scale ranging from 0 (none) to 3 (severe); Higher score indicates worse outcome. TOSS ranges from 0 (none) to 6 (severe): sum of 2 eye symptoms graded on a Likert scale each ranging from 0 (none) to 3 (severe) for itching/redness/gritty feeling & tearing/watering; Higher score indicates worse outcome. TSS ranges from 0 (none) to 18 (severe): sum of TNSS & TOSS combined; Higher score indicates worse outcome.
Time Frame: Day 190 from randomization (In-season); Timing may vary based on local season
Population: The "Number of Participants Analyzed" is the number of participants who received a second dose of the study drug. The "Number Analyzed" for each scale is the number of participants with available observed data for that scale.
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 38 | 33 | 37 | 38
Scores on a Scale
  TNSS | 4.49 (0.497) | 4.41 (0.520) | 5.07 (0.497) | 6.69 (0.469)
  TOSS | 1.90 (0.246) | 1.85 (0.257) | 1.83 (0.245) | 2.68 (0.232)
  TSS | 6.39 (0.692) | 6.26 (0.724) | 6.92 (0.690) | 9.36 (0.653)

30. Secondary Outcome: Daily Averaged TNSS, TOSS, TSS, Daily Medication Score (DMS) and Combined Symptom and Medication Score (CSMS) During Birch Pollen Season (BPS)
Description: TNSS ranges from 0 (none) to 12 (severe): Sum of 4 nasal symptoms (nasal congestion, itching, & runny nose, & sneezing) graded on a Likert scale from 0 (none) to 3 (severe); Higher score indicates worse outcome. TOSS ranges from 0 (none) to 6 (severe): Sum of 2 eye symptoms graded on Likert scale each from 0 (none) to 3 (severe) for itching/redness/gritty feeling & tearing/watering; Higher score indicates worse outcome. TSS ranges from 0 (none) to 18 (severe): Sum of TNSS & TOSS; Higher score indicates worse outcome. DMS ranges from 0 to 20 (max points): Sum for each pre-specified medication taken as oral antihistamine 6 points/dose (max daily score 6), ocular antihistamine 1.5 points/drop (max daily score 6), intranasal corticosteroid 2.0 points/spray (max daily score 8). CSMS ranges from 0 to 38 (max): Sum of DMS & TSS higher score indicates worse outcome). Daily TNSS, TOSS, TSS, DMS & CSMS each averaged over duration of birch pollen season presented.
Time Frame: Up to 253 days from randomization (during BPS)
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 38 | 33 | 39 | 39
Scores on a Scale
  TNSS | 3.38 (0.422) | 3.44 (0.443) | 3.57 (0.413) | 4.05 (0.399)
  TOSS | 1.09 (0.199) | 1.15 (0.210) | 1.16 (0.195) | 1.62 (0.188)
  TSS | 4.48 (0.595) | 4.59 (0.625) | 4.73 (0.582) | 5.65 (0.563)
  DMS | 0.84 (0.439) | 0.89 (0.457) | 1.05 (0.426) | 1.74 (0.408)
  CSMS | 5.350 (0.8912) | 5.509 (0.9352) | 5.776 (0.8710) | 7.392 (0.8433)

31. Secondary Outcome: Daily Averaged TNSS, TOSS, TSS, DMS and CSMS During Peak BPS
Description: TNSS ranges from 0 (none) to 12 (severe): Sum of 4 nasal symptoms (nasal congestion, itching, & runny nose, & sneezing) graded on a Likert scale from 0 (none) to 3 (severe); Higher score indicates worse outcome. TOSS ranges from 0 (none) to 6 (severe): Sum of 2 eye symptoms graded on Likert scale each from 0 (none) to 3 (severe) for itching/redness/gritty feeling & tearing/watering; Higher score indicates worse outcome. TSS ranges from 0 (none) to 18 (severe): Sum of TNSS & TOSS; Higher score indicates worse outcome. DMS ranges from 0 to 20 (max points): Sum for each pre-specified medication taken as oral antihistamine 6 points/dose (max daily score 6), ocular antihistamine 1.5 points/drop (max daily score 6), intranasal corticosteroid 2.0 points/spray (max daily score 8). CSMS ranges from 0 to 38 (max): Sum of DMS & TSS higher score indicates worse outcome). Daily TNSS, TOSS, TSS, DMS & CSMS each averaged over duration of peak birch pollen season presented.
Time Frame: Up to 253 days from randomization (during peak BPS)
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 37 | 33 | 39 | 39
Scores on a Scale
  TNNS | 3.79 (0.483) | 3.87 (0.502) | 3.71 (0.469) | 4.67 (0.452)
  TOSS | 1.24 (0.230) | 1.32 (0.238) | 1.25 (0.223) | 1.87 (0.214)
  TSS | 5.03 (0.679) | 5.18 (0.705) | 4.96 (0.659) | 6.53 (0.635)
  DMS | 0.94 (0.504) | 1.18 (0.517) | 1.11 (0.485) | 1.99 (0.463)
  CSMS | 5.997 (1.0154) | 6.357 (1.0525) | 6.055 (0.9842) | 8.501 (0.9500)

32. Secondary Outcome: Change From Pre-treatment Baseline in TNSS, TOSS, TSS, DMS and CSMS Averaged During BPS
Description: TNSS ranges from 0 (none) to 12 (severe): Sum of 4 nasal symptoms (nasal congestion, itching, & runny nose, & sneezing) graded on a Likert scale from 0 (none) to 3 (severe); Higher score indicates worse outcome. TOSS ranges from 0 (none) to 6 (severe): Sum of 2 eye symptoms graded on Likert scale each from 0 (none) to 3 (severe) for itching/redness/gritty feeling & tearing/watering; Higher score indicates worse outcome. TSS ranges from 0 (none) to 18 (severe): Sum of TNSS & TOSS; Higher score indicates worse outcome. DMS ranges from 0 to 20 (max points): Sum for pre-specified medication taken as oral antihistamine 6 points/dose (max daily score 6), ocular antihistamine 1.5 points/drop (max daily score 6), intranasal corticosteroid 2.0 points/spray (max daily score 8). CSMS ranges from 0 to 38 (max): Sum of DMS & TSS; Higher score indicates worse outcome. Change from pre-treatment baseline in TNSS, TOSS, TSS, DMS & CSMS each averaged over duration of birch pollen season presented.
Time Frame: Up to 253 days from randomization (during BPS)
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 38 | 33 | 39 | 39
Scores on a Scale
  TNSS | 1.38 (0.422) | 1.44 (0.443) | 1.57 (0.413) | 2.05 (0.399)
  TOSS | 0.54 (0.199) | 0.60 (0.210) | 0.61 (0.195) | 1.06 (0.188)
  TSS | 1.93 (0.595) | 2.03 (0.625) | 2.18 (0.582) | 3.10 (0.563)
  DMS | 0.78 (0.439) | 0.83 (0.457) | 0.98 (0.426) | 1.68 (0.408)
  CSMS | 2.733 (0.8912) | 2.891 (0.9352) | 3.158 (0.8710) | 4.775 (0.8433)

33. Secondary Outcome: Change From Pre-treatment Baseline in TNSS, TOSS, TSS, DMS and CSMS Averaged During Peak BPS
Description: TNSS ranges from 0 (none) to 12 (severe): Sum of 4 nasal symptoms (nasal congestion, itching, & runny nose, & sneezing) graded on Likert scale from 0 (none) to 3 (severe); Higher score indicates worse outcome. TOSS ranges from 0 (none) to 6 (severe): Sum of 2 eye symptoms graded on Likert scale each from 0 (none) to 3 (severe) for itching/redness/gritty feeling & tearing/watering; Higher score indicates worse outcome. TSS ranges from 0 (none) to 18 (severe): Sum of TNSS & TOSS; Higher score indicates worse outcome. DMS ranges from 0 to 20 (max points): Sum for pre-specified medication taken as oral antihistamine 6 points/dose (max daily score 6), ocular antihistamine 1.5 points/drop (max daily score 6), intranasal corticosteroid 2.0 points/spray (max daily score 8). CSMS ranges from 0 to 38 (max): Sum of DMS & TSS; Higher score indicates worse outcome. Change from pre-treatment baseline in TNSS, TOSS, TSS, DMS & CSMS each averaged over duration of peak birch pollen season presented.
Time Frame: Up to 253 days from randomization (during peak BPS)
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 37 | 33 | 39 | 39
Scores on a Scale
  TNSS | 1.79 (0.483) | 1.86 (0.502) | 1.71 (0.469) | 2.66 (0.452)
  TOSS | 0.69 (0.230) | 0.77 (0.238) | 0.70 (0.223) | 1.32 (0.214)
  TSS | 2.48 (0.679) | 2.62 (0.705) | 2.40 (0.659) | 3.97 (0.635)
  DMS | 0.88 (0.504) | 1.11 (0.517) | 1.04 (0.485) | 1.93 (0.463)
  CSMS | 3.376 (1.0154) | 3.736 (1.0525) | 3.434 (0.9842) | 5.880 (0.9500)

34. Secondary Outcome: Percent Change From Pre-treatment Baseline in TNSS, TOSS, TSS, DMS and CSMS Averaged During BPS
Description: TNSS range from 0 (none) to 12 (severe): Sum of 4 nasal symptoms (nasal congestion, itching, & runny nose, & sneezing) graded on Likert scale from 0 (none) to 3 (severe); Higher score indicates worse outcome. TOSS range from 0 (none) to 6 (severe): Sum of 2 eye symptoms graded on Likert scale each from 0 (none) to 3 (severe) for itching/redness/gritty feeling & tearing/watering; Higher score indicates worse outcome. TSS range from 0 (none) to 18 (severe): Sum of TNSS & TOSS; Higher score indicates worse outcome. DMS range from 0 to 20 (max points): Sum for pre-specified medication taken as oral antihistamine 6 points/dose (max daily score 6), ocular antihistamine 1.5 points/drop (max daily score 6), intranasal corticosteroid 2.0 points/spray (max daily score 8). CSMS range from 0 to 38 (max): Sum of DMS & TSS; Higher score indicates worse outcome. Percent change from pre-treatment baseline in TNSS, TOSS, TSS, DMS & CSMS each averaged over duration of birch pollen season presented.
Time Frame: Up to 253 days from randomization (during BPS)
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: Percentage of Change
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 38 | 33 | 39 | 39
Percentage of Change
  TNSS | 86.55 (32.120) | 81.60 (33.741) | 112.71 (31.414) | 120.74 (30.384)
  TOSS | -2.85 (18.480) | -0.66 (19.426) | 2.78 (18.078) | 44.16 (17.452)
  TSS | 126.46 (42.830) | 128.85 (45.018) | 147.59 (41.886) | 177.04 (40.526)
  DMS | -17.06 (43.686) | -15.13 (45.431) | 2.66 (42.367) | 70.85 (40.614)
  CSMS | 147.47 (65.846) | 187.32 (69.092) | 219.64 (64.352) | 263.58 (62.302)

35. Secondary Outcome: Percent Change From Pre-treatment Baseline in TNSS, TOSS, TSS, DMS and CSMS Averaged During Peak BPS
Description: TNSS range from 0 (none) to 12 (severe): Sum of 4 nasal symptoms (nasal congestion, itching, & runny nose, & sneezing) graded on Likert scale from 0 (none) to 3 (severe);Higher score indicates worse outcome. TOSS range from 0 (none) to 6 (severe): Sum of 2 eye symptoms graded on Likert scale each from 0 (none) to 3 (severe) for itching/redness/gritty feeling & tearing/watering;Higher score indicates worse outcome. TSS range from 0 (none) to 18 (severe): Sum of TNSS & TOSS;Higher score indicates worse outcome. DMS range from 0 to 20 (max points): Sum for pre-specified medication taken as oral antihistamine 6 points/dose (max daily score 6), ocular antihistamine 1.5 points/drop (max daily score 6), intranasal corticosteroid 2.0 points/spray (max daily score 8). CSMS range from 0 to 38 (max): Sum of DMS & TSS;Higher score indicates worse outcome. Percent change from pre-treatment baseline in TNSS, TOSS, TSS, DMS & CSMS each averaged over duration of peak birch pollen season presented.
Time Frame: Up to 253 days from randomization (during peak BPS)
Population: as for outcome 29
Measure: Least Squares Mean (Standard Error); unit: Percentage of Change
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 37 | 33 | 39 | 39
Percentage of Change
  TNSS | 103.41 (36.254) | 110.33 (37.612) | 121.50 (35.160) | 166.54 (33.905)
  TOSS | 9.74 (21.416) | 14.03 (22.233) | 10.21 (20.773) | 68.18 (19.993)
  TSS | 143.52 (48.745) | 165.35 (50.606) | 157.81 (47.273) | 234.84 (45.601)
  DMS | -7.34 (50.188) | 13.02 (51.510) | 8.63 (48.254) | 95.84 (46.109)
  CSMS | 164.04 (76.371) | 246.04 (79.156) | 227.73 (74.021) | 340.82 (71.451)

36. Secondary Outcome: Standardized Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ[S]) Score Averaged During BPS
Description: The RQLQ(S) is a self-administered questionnaire to measure health-related quality of life in those 12 years of age and above, as a result of perennial or seasonal allergic rhinitis. There are 28 items in 7 domains: activity limitation, sleep problems, nasal symptoms, eye symptoms, non-nasal/eye symptoms, practical problems, and emotional function with responses based on a 7-point Likert scale ranging from 0 (not troubled) to 6 (extremely troubled). Overall RQLQ(S) score is the mean of all 28 responses and the individual domain scores are the means of the items in those domains. Higher scores indicate more health-related quality of life impairment (lower scores are better). Overall RQLQ(S) score averaged over duration of birch pollen season presented.
Time Frame: Up to 253 days from randomization (during BPS)
Population: Randomized participants who received a second dose of the study drug
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 38 | 33 | 39 | 39
Scores on a Scale | 0.98 (0.205) | 0.98 (0.215) | 1.11 (0.197) | 1.29 (0.189)

37. Secondary Outcome: Standardized RQLQ(S) Score Averaged During Peak BPS
Description: The RQLQ(S) is a self-administered questionnaire to measure health-related quality of life in those 12 years of age and above, as a result of perennial or seasonal allergic rhinitis. There are 28 items in 7 domains: activity limitation, sleep problems, nasal symptoms, eye symptoms, non-nasal/eye symptoms, practical problems, and emotional function with responses based on a 7-point Likert scale ranging from 0 (not troubled) to 6 (extremely troubled). Overall RQLQ(S) score is the mean of all 28 responses and the individual domain scores are the means of the items in those domains. Higher scores indicate more health-related quality of life impairment (lower scores are better). Overall RQLQ(S) score averaged over duration of peak birch pollen season presented.
Time Frame: Up to 253 days from randomization (during peak BPS)
Population: Randomized participants who received a second dose of the study drug
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 38 | 33 | 39 | 39
Scores on a Scale | 1.04 (0.229) | 1.14 (0.239) | 1.25 (0.220) | 1.62 (0.215)

38. Secondary Outcome: Change From Pre-treatment Baseline in the Average RQLQ(S) Score During BPS
Description: The RQLQ(S) is a self-administered questionnaire to measure health-related quality of life in those 12 years of age and above, as a result of perennial or seasonal allergic rhinitis. There are 28 items in 7 domains: activity limitation, sleep problems, nasal symptoms, eye symptoms, non-nasal/eye symptoms, practical problems, and emotional function with responses based on a 7-point Likert scale ranging from 0 (not troubled) to 6 (extremely troubled). Overall RQLQ(S) score is the mean of all 28 responses and the individual domain scores are the means of the items in those domains. Higher scores indicate more health-related quality of life impairment (lower scores are better). Change from pre-treatment baseline averaged over duration of birch pollen season presented.
Time Frame: Up to 253 days from randomization (during BPS)
Population: Randomized participants who received a second dose of the study drug
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 37 | 32 | 39 | 39
Scores on a Scale | -0.11 (0.205) | -0.11 (0.215) | 0.02 (0.197) | 0.20 (0.189)

39. Secondary Outcome: Change From Pre-treatment Baseline in the Average RQLQ(S) Score During Peak BPS
Description: The RQLQ(S) is a self-administered questionnaire to measure health-related quality of life in those 12 years of age and above, as a result of perennial or seasonal allergic rhinitis. There are 28 items in 7 domains: activity limitation, sleep problems, nasal symptoms, eye symptoms, non-nasal/eye symptoms, practical problems, and emotional function with responses based on a 7-point Likert scale ranging from 0 (not troubled) to 6 (extremely troubled). Overall RQLQ(S) score is the mean of all 28 responses and the individual domain scores are the means of the items in those domains. Higher scores indicate more health-related quality of life impairment (lower scores are better). Change from pre-treatment baseline averaged over duration of peak birch pollen season presented.
Time Frame: Up to 253 days from randomization (during peak BPS)
Population: Randomized participants who received a second dose of the study drug
Measure: Least Squares Mean (Standard Error); unit: Scores on a Scale
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 36 | 32 | 39 | 38
Scores on a Scale | -0.04 (0.229) | 0.05 (0.239) | 0.16 (0.220) | 0.54 (0.215)

40. Secondary Outcome: Percent Change From Pre-treatment Baseline in the Average RQLQ(S) Score During BPS
Description: The RQLQ(S) is a self-administered questionnaire to measure health-related quality of life in those 12 years of age and above, as a result of perennial or seasonal allergic rhinitis. There are 28 items in 7 domains: activity limitation, sleep problems, nasal symptoms, eye symptoms, non-nasal/eye symptoms, practical problems, and emotional function with responses based on a 7-point Likert scale ranging from 0 (not troubled) to 6 (extremely troubled). Overall RQLQ(S) score is the mean of all 28 responses and the individual domain scores are the means of the items in those domains. Higher scores indicate more health-related quality of life impairment (lower scores are better). Percent change from pre-treatment baseline averaged over duration of birch pollen season presented.
Time Frame: Up to 253 days from randomization (during BPS)
Population: Randomized participants who received a second dose of the study drug
Measure: Least Squares Mean (Standard Error); unit: Percentage of Change
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 37 | 32 | 39 | 39
Percentage of Change | -32.68 (16.904) | -22.84 (17.780) | -12.70 (16.298) | 2.06 (15.598)

41. Secondary Outcome: Percent Change From Pre-treatment Baseline in the Average RQLQ(S) Score During Peak BPS
Description: The RQLQ(S) is a self-administered questionnaire to measure health-related quality of life in those 12 years of age and above, as a result of perennial or seasonal allergic rhinitis. There are 28 items in 7 domains: activity limitation, sleep problems, nasal symptoms, eye symptoms, non-nasal/eye symptoms, practical problems, and emotional function with responses based on a 7-point Likert scale ranging from 0 (not troubled) to 6 (extremely troubled). Overall RQLQ(S) score is the mean of all 28 responses and the individual domain scores are the means of the items in those domains. Higher scores indicate more health-related quality of life impairment (lower scores are better). Percent change from pre-treatment baseline averaged over duration of peak birch pollen season presented.
Time Frame: Up to 253 days from randomization (during peak BPS)
Population: Randomized participants who received a second dose of the study drug
Measure: Least Squares Mean (Standard Error); unit: Percentage of Change
Arm/Group | REGN5713-5714-5715 900 mg | REGN5713-5715 600 mg | REGN5715 300 mg | Placebo
Number analyzed (Participants) | 36 | 32 | 39 | 38
Percentage of Change | -27.67 (19.220) | -9.90 (20.000) | -1.67 (18.446) | 29.24 (17.972)

42. Secondary Outcome: Number of Participants With Any Treatment-Emergent Adverse Event (TEAE) Over the Study Duration
Time Frame: Up to 253 Days
Population: Randomized participants who receive any study drug, regardless of the amount of treatment administered
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | REGN5715 300 mg | REGN5713-5715 600 mg | REGN5713-5714-5715 900 mg
Number analyzed (Participants) | 55 | 55 | 51 | 55
Participants | 26 | 23 | 23 | 25

43. Secondary Outcome: Number of Participants With Any Treatment-Emergent Serious AE (TESAE) Over the Study Duration
Time Frame: Up to 253 Days
Population: Randomized participants who receive any study drug, regardless of the amount of treatment administered
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | REGN5715 300 mg | REGN5713-5715 600 mg | REGN5713-5714-5715 900 mg
Number analyzed (Participants) | 55 | 55 | 51 | 55
Participants | 0 | 0 | 0 | 0

44. Secondary Outcome: Serum Concentration of REGN5713 Over the Study Duration
Time Frame: Up to Week 36
Population: Randomized and treated participants who received REGN5713 and contributed to each timepoint
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | REGN5715 300 mg | REGN5713-5715 600 mg | REGN5713-5714-5715 900 mg
Number analyzed (Participants) | 0 | 45 | 54
mg/L
  Baseline |  | 0 (0) | 0 (0)
  Week 4: number analyzed (Participants) | 0 | 41 | 53
  Week 4 |  | 15.2 (4.72) | 16.2 (5.23)
  Week 8: number analyzed (Participants) | 0 | 40 | 43
  Week 8 |  | 7.10 (2.69) | 8.12 (3.59)
  Week 12: number analyzed (Participants) | 0 | 38 | 37
  Week 12 |  | 4.72 (2.37) | 5.25 (3.09)
  Week 18: number analyzed (Participants) | 0 | 31 | 34
  Week 18 |  | 2.18 (1.80) | 2.84 (2.60)
  Week 22: number analyzed (Participants) | 0 | 33 | 38
  Week 22 |  | 1.42 (1.27) | 2.04 (2.36)
  Week 27: number analyzed (Participants) | 0 | 33 | 38
  Week 27 |  | 16.9 (5.54) | 20.8 (8.40)
  Week 32: number analyzed (Participants) | 0 | 15 | 28
  Week 32 |  | 6.11 (3.10) | 6.52 (3.56)
  Week 36: number analyzed (Participants) | 0 | 33 | 38
  Week 36 |  | 2.88 (1.47) | 4.18 (3.02)

45. Secondary Outcome: Serum Concentration of REGN5714 Over the Study Duration
Time Frame: Up to Week 36
Population: Randomized and treated participants who received REGN5714 and contributed to each timepoint
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | REGN5715 300 mg | REGN5713-5715 600 mg | REGN5713-5714-5715 900 mg
Number analyzed (Participants) | 0 | 0 | 54
mg/L
  Baseline |  |  | 0 (0)
  Week 4: number analyzed (Participants) | 0 | 0 | 53
  Week 4 |  |  | 22.3 (5.96)
  Week 8: number analyzed (Participants) | 0 | 0 | 43
  Week 8 |  |  | 13.1 (4.36)
  Week 12: number analyzed (Participants) | 0 | 0 | 37
  Week 12 |  |  | 9.01 (3.70)
  Week 18: number analyzed (Participants) | 0 | 0 | 34
  Week 18 |  |  | 5.34 (3.69)
  Week 22: number analyzed (Participants) | 0 | 0 | 38
  Week 22 |  |  | 3.95 (3.45)
  Week 27: number analyzed (Participants) | 0 | 0 | 38
  Week 27 |  |  | 29.0 (9.51)
  Week 32: number analyzed (Participants) | 0 | 0 | 28
  Week 32 |  |  | 11.9 (4.92)
  Week 36: number analyzed (Participants) | 0 | 0 | 38
  Week 36 |  |  | 7.90 (4.10)

46. Secondary Outcome: Serum Concentration of REGN5715 Over the Study Duration
Time Frame: Up to Week 36
Population: Randomized and treated participants who received REGN5715 and contributed to each timepoint
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | REGN5715 300 mg | REGN5713-5715 600 mg | REGN5713-5714-5715 900 mg
Number analyzed (Participants) | 50 | 45 | 54
mg/L
  Baseline | 0 (0) | 0 (0) | 0 (0)
  Week 4: number analyzed (Participants) | 49 | 41 | 53
  Week 4 | 20.6 (5.94) | 21.5 (5.54) | 26.7 (9.37)
  Week 8: number analyzed (Participants) | 44 | 40 | 43
  Week 8 | 11.1 (3.35) | 12.3 (3.63) | 14.8 (4.96)
  Week 12: number analyzed (Participants) | 40 | 38 | 37
  Week 12 | 8.30 (3.42) | 8.73 (3.38) | 10.4 (4.28)
  Week 18: number analyzed (Participants) | 38 | 31 | 34
  Week 18 | 4.75 (3.27) | 4.51 (2.86) | 5.92 (4.17)
  Week 22: number analyzed (Participants) | 39 | 33 | 38
  Week 22 | 3.02 (2.20) | 3.12 (2.16) | 4.29 (3.77)
  Week 27: number analyzed (Participants) | 39 | 33 | 38
  Week 27 | 22.7 (8.40) | 24.4 (6.95) | 29.3 (9.29)
  Week 32: number analyzed (Participants) | 22 | 15 | 28
  Week 32 | 9.60 (4.09) | 10.7 (4.26) | 12.2 (4.93)
  Week 36: number analyzed (Participants) | 39 | 33 | 38
  Week 36 | 5.83 (2.42) | 6.16 (2.10) | 8.21 (4.21)

47. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) to REGN5713 Over Time
Time Frame: Up to Week 36
Population: Randomized and treated participants who received REGN5713 during the study
Measure: Count of Participants; unit: Participants
Arm/Group | REGN5715 300 mg | REGN5713-5715 600 mg | REGN5713-5714-5715 900 mg
Number analyzed (Participants) | 0 | 51 | 54
Participants
  Negative |  | 51 | 54
  Low Titer (<1000) Treatment Emergent Response |  | 0 | 0
  Moderate Titer (1000 to 10000) Treatment Emergent Response |  | 0 | 0
  High Titer (>10000) Treatment Emergent Response |  | 0 | 0

48. Secondary Outcome: Number of Participants With ADA to REGN5714 Over Time
Time Frame: Up to Week 36
Population: Randomized and treated participants who received REGN5714 during the study
Measure: Count of Participants; unit: Participants
Arm/Group | REGN5715 300 mg | REGN5713-5715 600 mg | REGN5713-5714-5715 900 mg
Number analyzed (Participants) | 0 | 0 | 54
Participants
  Negative |  |  | 53
  Low Titer (<1000) Treatment Emergent Response |  |  | 1
  Moderate Titer (1000 to 10000) Treatment Emergent Response |  |  | 0
  High Titer (>10000) Treatment Emergent Response |  |  | 0

49. Secondary Outcome: Number of Participants With ADA to REGN5715 Over Time
Time Frame: Up to Week 36
Population: Randomized and treated participants who received REGN5715 during the study
Measure: Count of Participants; unit: Participants
Arm/Group | REGN5715 300 mg | REGN5713-5715 600 mg | REGN5713-5714-5715 900 mg
Number analyzed (Participants) | 54 | 51 | 54
Participants
  Negative | 53 | 50 | 53
  Low Titer (<1000) Treatment Emergent Response | 1 | 1 | 1
  Moderate Titer (1000 to 10000) Treatment Emergent Response | 0 | 0 | 0
  High Titer (>10000) Treatment Emergent Response | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time of signing the informed consent form (ICF) up to Day 260
Arm/Group | Placebo | REGN5715 300 mg | REGN5713-5715 600 mg | REGN5713-5714-5715 900 mg
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55 | 0/51 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55 | 0/51 | 0/55
Other Adverse Events (participants affected / at risk) | 23/55 | 19/55 | 20/51 | 19/55
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=55) | REGN5715 300 mg (N=55) | REGN5713-5715 600 mg (N=51) | REGN5713-5714-5715 900 mg (N=55)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 8 (8) | 5 (7) | 3 (5)
COVID-19 (Infections and infestations) | 4 (4) | 3 (3) | 5 (5) | 2 (2)
Headache (Nervous system disorders) | 8 (16) | 4 (7) | 10 (17) | 7 (8)
Presyncope (Nervous system disorders) | 3 (3) | 3 (3) | 2 (2) | 2 (3)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 1 (2) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 1 (1) | 4 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (6)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (2)
Injection site erythema (General disorders) | 2 (7) | 1 (1) | 4 (6) | 2 (3)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Injection site pruritus (General disorders) | 3 (8) | 0 (0) | 3 (3) | 1 (1)
Hepatic enzyme increased (Investigations) | 3 (3) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the Sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT05430919/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT05430919/SAP_001.pdf